CLINICAL TRIAL: NCT06349252
Title: Survival Validation and Gene Mutations of N Descriptors in the Ninth Edition of the TNM Classification for Lung Cancer
Status: Recruiting | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Haiquan Chen, The director of the department of thoracic surgery, Fudan University
Other Study IDs: LUNGTNM
Record Dates: First submitted 2024-03-31; First posted 2024-04-05 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-03

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Radical resection — Patients should undergo radical resection.

SUMMARY:
The International Association for the Study of Lung Cancer Staging Committee recently unveiled the ninth edition of TNM staging system for lung cancer. This study aims to explore survival outcomes, stage grouping, and gene mutations in N descriptors of this new classification system.

ELIGIBILITY:
Inclusion Criteria:

Pathological N2.

Exclusion Criteria:

Patients undergoing neoadjuvant chemotherapy

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with pathological N2 non-small cell lung cancer based on the eighth TNM staging system in Fudan University Shanghai Cancer Center.
Sampling Method: Probability Sample
Enrollment: 1263 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | Five year

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Cancer Center, Shanghai, Shanghai Municipality, China